CLINICAL TRIAL: NCT05596916
Title: The Effect of Axio Scapular Muscle Stretching Exercises on Posture, Periscapular Muscle Strength and Disability in Office Workers
Brief Title: The Effect of Axio Scapular Muscle Stretching Exercises in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Kus, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MustafaKU06
Record Dates: First submitted 2022-10-18; First posted 2022-10-27 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Neck Muscle Issue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency of stretching exercise (Experimental): Axio scapular muscle stretching exercises will be applied for 5 days a week during 6 weeks
  Interventions: Other: High frequency of stretching exercise
- Low frequency of stretching exercise (Active Comparator): Axio scapular muscle stretching exercises will be applied for 3 days a week during 6 weeks
  Interventions: Other: Low frequency of stretching exercise

INTERVENTIONS:
Other: High frequency of stretching exercise — After the randomization and evaluations, the selected postural stretching exercises will be taught to both groups in the clinic, and then a brochure will be given to the participants and they will be asked to practice these exercises at home.
  In the experimental group, the exercises will be applied at the specified time and frequency, 5 days a week.
  Participants will be given an "Exercise Diary" and exercise tracking will be provided by calling the participants once a week. The exercises will be done for 6 weeks. Participants will be evaluated twice, before and end of the treatment.
  Arms: High frequency of stretching exercise
Other: Low frequency of stretching exercise — After the randomization and evaluations, the selected postural stretching exercises will be taught to both groups in the clinic, and then a brochure will be given to the participants and they will be asked to practice these exercises at home.
  In the experimental group, the exercises will be applied at the specified time and frequency, 3 days a week.
  Participants will be given an "Exercise Diary" and exercise tracking will be provided by calling the participants once a week. The exercises will be done for 6 weeks. Participants will be evaluated twice, before and end of the treatment.
  Arms: Low frequency of stretching exercise

SUMMARY:
The aim of this study is to examine the effects of stretching exercises applied to the axioscapular muscles on posture, periscapular muscle strength and symptoms in office workers.

DETAILED DESCRIPTION:
Individuals who work at a desk for a long time often take a kyphotic or loose sitting position, resulting in tension in some of the axioscapular muscles and weakness in others. Because, as a result of wrong working posture at the desk, scapular downward rotation formation, increased activation in trapezius and levator scapula muscles, pain, decrease in normal joint range of motion (ROM) may result in impaired proprioception and this situation may create a vicious circle. In addition, incorrect sitting posture was found to be associated with changes in scapula position, kinematics and muscle activity.

It is considered a clinical feature that a change in scapular alignment can cause neck pain and dysfunction. The scapula shares common muscle connections with the neck, and altered axioscapular muscle function is claimed to potentially cause neck pain through abnormal loading of the cervical spine or the formation of myofascial trigger points.

Stretching the shortened upper trapezius, sternocleidomastoid, and levator scapula muscles and strengthening the deep cervical flexor muscles are effective in correcting the anterior tilt posture of the head.

Stretching exercises applied to the tension and shortness of the axioscapular muscles can have a positive effect on middle and lower trapezius muscle and serratus anterior muscle weakness, as they contribute to the change of scapular position. It may also contribute to cervical motion and/or symptom relief.

For this reason, the aim of the study is to examine the effects of axioscapular muscle stretching exercises on posture, periscapular muscle strength and symptoms in office workers. In addition, information about the effect of isolated stretching exercises on muscle strength and symptoms will be obtained and a contribution will be made about the weekly dosage.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer office workers who work at a desk more than 4 hours a day for at least 1 year

Exclusion Criteria:

* Those who have undergone surgery on the upper extremity and/or neck,
* Patients that had been diagnosed for Diabetes, Rheumatoid Arthritis, Ankylosing Spondylitis,
* Those who have received a physiotherapy program for the neck and/or upper extremity in the last 3 months,
* People who are actively involved in sports (at least 3 days a week / 150 minutes).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
The anterior tilt of head analysis with photography method | Evaluations will be done between two time points: first time at baseline and second time after 6-weeks rehabilitation program.
  Markers will be placed on the ear tragus, C7 and T12 process prominences, and acromion, and sagittal plane photographs will be taken. The angle of the anterior tilt of the head will be evaluated through these photographs.
The shoulder protraction analysis with photography method | Evaluations will be done between two time points: first time at baseline and second time after 6-weeks rehabilitation program.
  Markers will be placed on the ear tragus, C7 and T12 process prominences, and acromion, and sagittal plane photographs will be taken. The angle of shoulder protraction will be evaluated through these photographs.
The thoracic kyphosis analysis with photography method | Evaluations will be done between two time points: first time at baseline and second time after 6-weeks rehabilitation program.
  Markers will be placed on the ear tragus, C7 and T12 process prominences, and acromion, and sagittal plane photographs will be taken. The angle of thoracic kyphosis will be evaluated through these photographs.
Shoulder protraction with tape measure | Evaluations will be done between two time points: first time at baseline and second time after 6-weeks rehabilitation program.
  In addition, shoulder protraction with tape measure; It will be evaluated by measuring the distance between the acromion and the bed, with the person lying on his back.
The hand held dynamometer | Evaluations will be done between two time points: first time at baseline and second time after 6-weeks rehabilitation program.
  Muscle strength (Lower and Middle Trapezius Muscles, Serratus Anterior) will be evaluated with a hand held dynamometer. The selected muscles will be tested to achieve a maximum isometric contraction of 3 repetitions in the appropriate anatomical position.

SECONDARY OUTCOMES:
Quick DASH (Disabilities of the Arm, Shoulder and Hand) Questionnaire | Evaluations will be done between two time points: first time at baseline and second time after 6-weeks rehabilitation program.
  Quick DASH is a 11-item questionnaire that questions the activities of a person in daily life, the degree of participation in recreational activities, the symptom and psychosocial state that affects their pain, and sleep quality. The total score is at least 0 and at most 100, and the high scores are positively correlated with the decreased functional level.
Modified Neck Disability Index | Evaluations will be done between two time points: first time at baseline and second time after 6-weeks rehabilitation program.
  This form consists of 10 questions. The intensity of pain in the neck, difficulty in personal care, ability to lift weights, the interaction of reading with neck pain, headaches, difficulty in doing work, difficulty in driving, sleeping and leisure activities are questioned. Each question scores between 0 and 5 points, and an increased score is associated with increased disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Hatay, Alahan, Turkey (Türkiye)